CLINICAL TRIAL: NCT01154699
Title: Positive Airway Pressure for the Treatment of Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Robert L. Owens, Instructor in Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2009-P-001733/1; 1F32HL097578-01 (NIH); 5K23HL105542 (NIH)
Record Dates: First submitted 2010-06-18; First posted 2010-07-01 (Estimated); Results first posted 2017-05-17 (Actual); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Asthma; Sleep Apnea
Keywords: Asthma; Nocturnal Asthma; Lung volumes; Deep inspiration; Obstructive sleep apnea
MeSH Terms: conditions — Asthma; Sleep Apnea Syndromes; Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care first, then Bilevel PAP (Experimental): Subjects will begin the study by continuing their usual care for 4 weeks. They will complete questionnaires and breathing tests at the start and end of this 4 week period. After a "Washout Period" of an additional 4 weeks of usual care, they will then start Bilevel PAP therapy for 4 weeks. Just before and after the Bilevel PAP they will complete questionnaires and breathing tests.
  Interventions: Device: Bilevel PAP (4 weeks); Other: Usual Care (4 weeks); Other: Washout Period (4 weeks)
- Bilevel PAP first, then Usual Care (Experimental): Subjects will begin the study by starting on Bilevel PAP for 4 weeks. Just before and after the Bilevel PAP they will complete questionnaires and breathing tests. After a 4 week "Washout Period" of usual care, they will start a Usual Care period for 4 weeks. They will complete questionnaires and breathing tests at the start and end of this 4 week period.
  Interventions: Device: Bilevel PAP (4 weeks); Other: Usual Care (4 weeks); Other: Washout Period (4 weeks)

INTERVENTIONS:
Device: Bilevel PAP (4 weeks) — Subjects will use bilevel PAP each night for 4 weeks. The pressure levels will be adjusted by the investigators to increase lung volumes during the night.
  Other Names: Bilevel positive airway pressure
Other: Usual Care (4 weeks) — Subjects will continue with their usual asthma care. Investigators will make no changes to their medications or other habits.
Other: Washout Period (4 weeks) — Subjects will continue with their usual asthma care in between the Usual Care and Bilevel PAP periods. Investigators will make no changes to their medications or other habits.

SUMMARY:
Asthma is an extremely common disorder, which is becoming more prevalent. The purpose of this study is to examine how nocturnal lung volumes contribute to asthma severity, which may explain part of the link between asthma and obesity. The investigators seek to test the hypothesis that raising lung volumes during the night will improve asthma symptoms. The investigators work may lead to new targets for therapy.

DETAILED DESCRIPTION:
Asthma is a chronic respiratory disease characterized by airway inflammation and airway hyperresponsiveness, which causes airflow obstruction. It is extremely prevalent, affecting an estimated 22 million Americans, and costly with loss of productivity and direct healthcare costs in the billions of dollars. The incidence and prevalence of asthma are increasing, both in the US and around the world. This increase comes despite greater understanding of the inflammatory and allergic basis for asthma, and despite better antiinflammatory medications. One explanation for the increasing prevalence of asthma is the concomitant increase in obesity, with the majority of Americans now overweight or obese. Numerous studies have convincingly linked asthma and obesity, and demonstrated increased obstruction with weight gain and decreased obstruction with weight loss. However, the mechanisms that underlie this linkage are not known.

We believe that low lung volumes contribute to the pathogenesis and severity of asthma. End-expiratory lung volume is decreased in obesity, and likely falls further during sleep, particularly in overweight and obese patients. Both upper and lower airway resistance increase with decreasing lung volumes, as airways become smaller. However, prior work has shown that lower airway resistance increases out of proportion to the decrease in lung volume that occurs during sleep in asthma patients. This difference between controls and people with asthma has not been further explored, yet may provide insight into asthma pathogenesis and provide potential targets for therapy.

Therefore, we propose a series of experiments to define the impact of lung volumes during sleep on airway resistance. One of these experiments will be to to test the hypothesis that lung stretch can be used therapeutically by tonically and dynamically increasing lung volumes during sleep using bi-level positive airway pressure. This research can help delineate asthma pathogenesis and may help improve therapeutic options in this exceedingly common disease.

ELIGIBILITY:
Inclusion Criteria:

* mild to moderate asthma, diagnosed by a physician, OR
* mild to moderate asthma and CPAP treated OSA. Must be compliant with CPAP therapy (greater than 4 hours per night, at least 4 nights/week)

Exclusion Criteria:

* lung disease other than asthma or OSA
* medications known to affect respiratory function (apart from asthma and rhinitis therapy)
* abnormal nasal anatomy
* current smokers and ex-smokers (quit within the last 3 months, or >10 pack-years)
* pregnant women - women of child bearing age will undergo a urine pregnancy test before enrollment and during the course of the study, as some of the study procedures cannot be performed during pregnancy and because pregnancy often changes asthma symptoms and severity.
* severe asthma - defined as a recent exacerbation (doctor or ER visit for asthma, or oral steroid use, within the previous 4 weeks) or frequent exacerbations (>4 exacerbations in the last year.
* severe obstructive sleep apnea requiring supplemental oxygen in addition to CPAP therapy.
* the regular use of prescription (e.g. zolpidem) or over-the-counter sleep aids (e.g. Benadryl).
* Central sleep apnea

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2010-07; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert L Owens, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 33 subjects were assessed for eligibility (20 asthma only, 13 asthma + OSA).
  12 were excluded, with 11 not meeting inclusion criteria, and 1 declining to participate.
Period: First Intervention (4 Weeks)
Arm/Group | Usual Care First, Then Bilevel PAP | Bilevel PAP First, Then Usual Care
Started | 13 | 8
Subjects With Asthma Only (The number of subjects who had asthma but NOT OSA in each arm) | 7 | 6
Subjects With Asthma + OSA (The number of subjects who had asthma and OSA in each arm) | 6 | 2
Completed | 13 | 8
Not Completed | 0 | 0
Period: Washout Period (4 Weeks)
Arm/Group | Usual Care First, Then Bilevel PAP | Bilevel PAP First, Then Usual Care
Started | 13 | 8
Subjects With Asthma Only | 7 | 6
Subjects With Asthma + OSA | 6 | 2
Completed | 13 | 8
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Usual Care First, Then Bilevel PAP | Bilevel PAP First, Then Usual Care
Started | 13 | 8
Subjects With Asthma Only | 7 | 6
Subjects With Asthma + OSA | 6 | 2
Completed | 13 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Asthma Only: Subjects meeting all inclusion criteria and no exclusion criteria with asthma only (no sleep apnea)
- Asthma + OSA: Subjects meeting all inclusion criteria and no exclusion criteria with asthma and obstructive sleep apnea on continuous positive airway pressure (CPAP) treatment
- Total: Total of all reporting groups
Arm/Group | Asthma Only | Asthma + OSA | Total
Number analyzed (Participants) | 13 | 8 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.2 (16.7) | 44.75 (10.5) | 43.8 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 5 | 14
  Male | 4 | 3 | 7
Region of Enrollment [Number; unit: participants]
  United States | 13 | 8 | 21
Body Mass Index (kg/m2) [Mean (Standard Deviation); unit: kg/m2] | 30.5 (7.4) | 36.4 (5.2) | 32.7 (7.2)
FEV1% predicted [Mean (Standard Deviation); unit: %] | 90.2 (21.3) | 89.4 (21.0) | 89.9 (20.7)
FEV1/FVC [Mean (Standard Deviation); unit: ratio] | 0.75 (0.09) | 0.75 (.06) | 0.75 (.07)
PC20 (mg/mL) [Geometric Mean (Standard Deviation); unit: mg/mL] | 1.5 (0.5) | 1.8 (1.4) | 1.6 (0.3)
AHI (events/hour) [Mean (Standard Deviation); unit: events per hour] | 2.5 (2.3) | 40.0 (30.1) | 11.6 (3.4)
CPAP Pressure [Mean (Standard Deviation); unit: cm of water] — Population: Subjects with ASTHMA only do not use CPAP
  cm of water
    number analyzed (Participants) | 0 | 8 | 8
    (all) |  | 11.6 (3.4) | 11.6 (3.4)
CPAP Usage [Mean (Standard Deviation); unit: minutes] — Population: Subjects with asthma ONLY do not use CPAP
  minutes
    number analyzed (Participants) | 0 | 8 | 8
    (all) |  | 264 (96) | 264 (96)

OUTCOME MEASURES:

1. Primary Outcome: Asthma Control Test
Description: Well validated questionnaire of asthma symptoms which includes 5 written questions. Each question is answered on a scale of 1-5, which are summed to report a range of asthma control from 5 to 25 (higher score indicates better asthma control).
Time Frame: Every 4 weeks during the 12 week study (at the start and end of the Usual Care period, and at the start and end of the Bilevel PAP intervention period)
Population: All 21 patients went through usual care and bilevel PAP therapy
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Usual Care: Subjects will begin the study by continuing their usual care for 4 weeks. They will complete questionnaires and breathing tests at the start and end of this 4 week period.
- Bilevel PAP: Subjects will wear Bilevel PAP for 4 weeks. Just before and after the Bilevel PAP they will complete questionnaires and breathing tests.
Arm/Group | Usual Care | Bilevel PAP
Number analyzed (Participants) | 21 | 21
units on a scale
  Pre | 19.3 (5.1) | 19.8 (3.4)
  Post | 19.1 (4.6) | 19.6 (4.2)
Statistical Analysis 1: Comparison: Usual Care vs Bilevel PAP; The difference in the change in asthma control during the Usual care and the Bilevel PAP period were compared; Test type: Superiority or Other; p = 0.8, t-test, 2 sided

2. Primary Outcome: Airway Reactivity as Measured by Methacholine Challenge (PC20)
Description: This is a physiological measurement derived from repeated breathing maneuvers which measures airway reactivity. Subjects are exposed to higher and higher concentrations of an airway irritant (in this case methacholine), and between each dose perform spirometry. The test is stopped after the forced expiratory volume in 1 second (FEV1) falls 20% below the baseline. The concentration of methacholine at which this occurs is called the PC20. Methacholine challenges are routinely used in the diagnosis of asthma, and in many asthma research studies to measure changes in airway reactivity.
Time Frame: as for outcome 1
Population: All subjects completed the crossover study design
Measure: Geometric Mean (Standard Error); unit: mg/mL
Groups:
- Usual Care: Subjects record asthma quality of life and symptoms, without intervention for 4 weeks.
- Bi-level PAP: Subjects wear Bi-level PAP during the night for 4 weeks, and record asthma quality of life and asthma symptoms.
  Bi-level positive airway pressure (bi-level PAP): Subjects will use bi-level PAP each night for 4 weeks. The pressure levels will be adjusted by the investigators to increase lung volumes during the night.
Arm/Group | Usual Care | Bi-level PAP
Number analyzed (Participants) | 21 | 21
mg/mL
  Pre | 1.3 (0.31) | 1.24 (1.97)
  Post | 0.88 (2.41) | 1.36 (2.13)
Statistical Analysis 1: Comparison: Usual Care vs Bi-level PAP; Change in PC20 between the two arms; Test type: Superiority or Other; p = 0.20, t-test, 2 sided

3. Secondary Outcome: Epworth Sleepiness Scale (ESS)
Description: 8 item questionnaire to measure daytime sleepiness, with total score reported 0 (less sleepy) to 24 (most sleepy). Scores greater than or equal to 10 are considered excessive daytime sleepiness.
Time Frame: as for outcome 1
Population: All subjects completed both arms of this crossover study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Bi-level PAP
Number analyzed (Participants) | 21 | 21
units on a scale
  Pre | 9.1 (5.4) | 9.8 (5.0)
  Post | 9.7 (4.6) | 9.1 (5.2)
Statistical Analysis 1: Comparison: Usual Care vs Bi-level PAP; Test type: Superiority or Other; p = 0.78, t-test, 2 sided

4. Secondary Outcome: Pittsburgh Sleep Quality Index (PSQI)
Description: Well validated questionnaire used frequently to measure sleep quality over the prior 1 month. It consists of 19 individual items that combine to form 7 components summed to create one global score. The overall score is between 0 (better sleep) and 21 (worse sleep).
Time Frame: as for outcome 1
Population: All subjects completed both arms of this crossover study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Bi-level PAP
Number analyzed (Participants) | 21 | 21
units on a scale
  pre | 6.8 (4.0) | 6.6 (3.3)
  post | 6.1 (3.4) | 6.1 (4.1)
Statistical Analysis 1: Comparison: Usual Care vs Bi-level PAP; Test type: Superiority or Other; p = 0.61, t-test, 2 sided

5. Secondary Outcome: Short Form (SF-36) Health Survey
Description: Well validated quality of life questionnaire that measures eight sub-sections, which are summed to yield a score from 0 (maximal disability) to 100 (no disability). The eight subsections are: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, mental health.
Time Frame: as for outcome 1
Population: All subjects completed both arms of the study
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Bi-level PAP
Number analyzed (Participants) | 21 | 21
units on a scale
  pre | 70.8 (15.4) | 74.0 (14.5)
  post | 70.3 (16.8) | 73.5 (16.6)
Statistical Analysis 1: Comparison: Usual Care vs Bi-level PAP; Test type: Superiority or Other; p = 0.94, t-test, 2 sided

6. Secondary Outcome: FEV1 %Predicted
Description: Performed as part of spirometry
Time Frame: as for outcome 1
Population: All subjects completed both arms of this crossover study.
Measure: Mean (Standard Deviation); unit: percentage of predicted FEV1
Arm/Group | Usual Care | Bi-level PAP
Number analyzed (Participants) | 21 | 21
percentage of predicted FEV1
  pre | 89.9 (20.7) | 87.1 (22.4)
  post | 88.1 (22.3) | 89.7 (20.0)
Statistical Analysis 1: Comparison: Usual Care vs Bi-level PAP; Test type: Superiority or Other; p = 0.76, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Asthma Only | Asthma + OSA
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/8
Other Adverse Events (participants affected / at risk) | 3/13 | 0/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Asthma Only (N=13) | Asthma + OSA (N=8)
Central Sleep Apnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) — Patients naive to PAP therapy developed central apneas while on bilevel PAP therapy

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No